CLINICAL TRIAL: NCT05284838
Title: The FAIL CT Study: Facilitating Adaptive Expertise in Learning Computed Tomography, a Multi-center Randomized Controlled Trial
Brief Title: Facilitating Adaptive Expertise in Learning Computed Tomography
Acronym: FAIL CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Brown University (Other); Alameda Health System (Other); University of California, Los Angeles (Other); University of Chicago (Other); The University of Texas Health Science Center, Houston (Other); University of Wisconsin, Madison (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Leonardo Aliaga, Clinical Instructor, Department of Emergency Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 64099
Record Dates: First submitted 2022-03-10; First posted 2022-03-17 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Adaptive Expertise; Error Management Training; Learning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Error Management Training (Difficult) (Experimental): Participants receive the learning strategy Error Management Training and encounter difficult questions.
  Interventions: Other: Error Management Training (Difficult)
- Error Management Training (Easy) (Experimental): Participants receive the learning strategy Error Management Training and encounter easy questions.
  Interventions: Other: Error Management Training (Easy)
- Error Avoidance Training (Active Comparator): Participants receive the learning strategy Error Avoidance Training.
  Interventions: Other: Error Avoidance Training

INTERVENTIONS:
Other: Error Management Training (Difficult) — Error Management Training is used to teach head computed tomography interpretation. Participants encounter difficult questions.
  Arms: Error Management Training (Difficult)
Other: Error Management Training (Easy) — Error Management Training is used to teach head computed tomography interpretation. Participants encounter easy questions.
  Arms: Error Management Training (Easy)
Other: Error Avoidance Training — Error Avoidance Training used to teach head computed tomography interpretation.
  Arms: Error Avoidance Training

SUMMARY:
The main objective of this study is to demonstrate that Error Management Training improves adaptive expertise in head computed tomography interpretation. The investigators will conduct a randomized controlled trial comparing two learning strategies, Error Management Training vs Error Avoidance Training, in emergency medicine residents. The investigators hypothesize that Error Management Training, as compared to Error Avoidance Training, will improve adaptive expertise, as measured by skills transfer, when used to teach head computed tomography interpretation to emergency medicine residents.

DETAILED DESCRIPTION:
Adaptive expertise is the ability to apply existing skills to novel situations. Adaptive expertise enables physicians to reduce preventable medical errors when managing clinical scenarios not encountered during training. However, residency curricula rarely address this learning outcome. Error Management Training improves transfer of skills to new contexts and develops adaptive expertise. Although this methodology has been shown to improve adaptive expertise in procedural skills, its impact on cognitive skills in medical training remains underexplored. Error Management Training promises to improve patient care by developing emergency physicians' adaptive expertise. However, the investigators need further evidence for its efficacy with cognitive skills in residency training. The investigators aim to demonstrate that Error Management Training improves adaptive expertise in a cognitive skill, using head computed tomography interpretation as a model.

ELIGIBILITY:
Inclusion Criteria:

* Study participation will be available to all current emergency medicine residents at Stanford and at thirteen external sites.

Exclusion Criteria:

* Adults unable to consent
* Pregnant women
* Individuals who are not yet adults (infants, children, teenagers)
* Prisoners
* Medical students
* Residents from specialties other than emergency medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Percent correct on an assessment of transfer of skills (adaptive expertise) | Immediately after instructional session (up to 60 minutes to complete the assessment)
  Participants will have to demonstrate transfer of head computed tomography interpretation skills by interpreting novel radiology cases different from those used in the instructional session. Performance will be assessed by percent score on a head computed tomography interpretation test using novel radiology content not addressed in the instructional session. Score range is 0-100%.

SECONDARY OUTCOMES:
Percent correct on an assessment of post-session proficiency for learning objectives (routine expertise) | Immediately after instructional session (up to 60 minutes to complete the assessment)
  Participants will have to demonstrate direct application of the intervention's learning objectives by interpreting radiology cases similar to those used in the instructional session. Performance will be assessed by percent score on a head computed tomography interpretation test using radiology content similar to that used in the instructional session. Score range is 0-100%.
Effect of post-graduate year level on post-test performance | Immediately after instructional session (up to 60 minutes to complete the assessment)
  Performance on a head computed tomography interpretation test (both adaptive expertise and routine expertise cases) will be assessed by percent score, stratified by post-graduate year level to show differences across residency training stage. Score range is 0-100%.
Mediation effect of errors on performance on the adaptive expertise cases | Number of errors will be measured during the educational intervention
  The number of errors made during the educational intervention will be measured for both the Error Management Training (Difficult) arm and the Error Management Training (Easy) arm. A mediation analysis will be conducted to assess the effect of committing errors during learning on subsequent performance in the cases measuring adaptive expertise.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Aliaga, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

REFERENCES:
- [Background] Aliaga L, Clarke SO. Rethinking Radiology: An Active Learning Curriculum for Head Computed Tomography Interpretation. West J Emerg Med. 2022 Jan 1;23(1):47-51. doi: 10.5811/westjem.2021.10.53665. PMID 35060860
- [Background] Pusic MV, Santen SA, Dekhtyar M, Poncelet AN, Roberts NK, Wilson-Delfosse AL, Cutrer WB. Learning to balance efficiency and innovation for optimal adaptive expertise. Med Teach. 2018 Aug;40(8):820-827. doi: 10.1080/0142159X.2018.1485887. Epub 2018 Aug 9. PMID 30091659
- [Background] Royce CS, Hayes MM, Schwartzstein RM. Teaching Critical Thinking: A Case for Instruction in Cognitive Biases to Reduce Diagnostic Errors and Improve Patient Safety. Acad Med. 2019 Feb;94(2):187-194. doi: 10.1097/ACM.0000000000002518. PMID 30398993
- [Background] King A, Holder MG Jr, Ahmed RA. Errors as allies: error management training in health professions education. BMJ Qual Saf. 2013 Jun;22(6):516-9. doi: 10.1136/bmjqs-2012-000945. Epub 2013 Jan 3. PMID 23293120
- [Background] Dyre L, Tabor A, Ringsted C, Tolsgaard MG. Imperfect practice makes perfect: error management training improves transfer of learning. Med Educ. 2017 Feb;51(2):196-206. doi: 10.1111/medu.13208. Epub 2016 Dec 12. PMID 27943372
- [Background] Gardner AK, Abdelfattah K, Wiersch J, Ahmed RA, Willis RE. Embracing Errors in Simulation-Based Training: The Effect of Error Training on Retention and Transfer of Central Venous Catheter Skills. J Surg Educ. 2015 Nov-Dec;72(6):e158-62. doi: 10.1016/j.jsurg.2015.08.002. Epub 2015 Sep 8. PMID 26362712
- [Background] Mylopoulos M, Brydges R, Woods NN, Manzone J, Schwartz DL. Preparation for future learning: a missing competency in health professions education? Med Educ. 2016 Jan;50(1):115-23. doi: 10.1111/medu.12893. PMID 26695471
- [Background] Keith N, Frese M. Effectiveness of error management training: a meta-analysis. J Appl Psychol. 2008 Jan;93(1):59-69. doi: 10.1037/0021-9010.93.1.59. PMID 18211135
- [Background] Keith N, Frese M. Self-regulation in error management training: emotion control and metacognition as mediators of performance effects. J Appl Psychol. 2005 Jul;90(4):677-91. doi: 10.1037/0021-9010.90.4.677. PMID 16060786
- [Background] Kua J, Lim WS, Teo W, Edwards RA. A scoping review of adaptive expertise in education. Med Teach. 2021 Mar;43(3):347-355. doi: 10.1080/0142159X.2020.1851020. Epub 2020 Nov 28. PMID 33251895
- [Background] Eva KW. Diagnostic error in medical education: where wrongs can make rights. Adv Health Sci Educ Theory Pract. 2009 Sep;14 Suppl 1:71-81. doi: 10.1007/s10459-009-9188-9. Epub 2009 Aug 11. PMID 19669913
- [Background] Soderstrom NC, Bjork RA. Learning versus performance: an integrative review. Perspect Psychol Sci. 2015 Mar;10(2):176-99. doi: 10.1177/1745691615569000. PMID 25910388
- [Background] Metcalfe J. Learning from Errors. Annu Rev Psychol. 2017 Jan 3;68:465-489. doi: 10.1146/annurev-psych-010416-044022. Epub 2016 Sep 14. PMID 27648988
- [Background] Mylopoulos M, Kulasegaram K, Woods NN. Developing the experts we need: Fostering adaptive expertise through education. J Eval Clin Pract. 2018 Jun;24(3):674-677. doi: 10.1111/jep.12905. Epub 2018 Mar 8. PMID 29516651
- [Background] Mylopoulos M, Steenhof N, Kaushal A, Woods NN. Twelve tips for designing curricula that support the development of adaptive expertise. Med Teach. 2018 Aug;40(8):850-854. doi: 10.1080/0142159X.2018.1484082. Epub 2018 Jul 15. PMID 30009648
- [Derived] Aliaga L, Bavolek RA, Cooper B, Mariorenzi A, Ahn J, Kraut A, Duong D, Burger C, Gisondi MA. Error Management Training and Adaptive Expertise in Learning Computed Tomography Interpretation: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2431600. doi: 10.1001/jamanetworkopen.2024.31600. PMID 39250155